CLINICAL TRIAL: NCT04852913
Title: Effects of Bowen's Technique In Postural Neck Pain Among Dentist
Brief Title: Bowen's Technique In Postural Neck Pain Among Dentist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00857 Nida Aslam
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Neck Pain
Keywords: Pain; Dentist; Neck; Bowen technique
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen's Technique (Experimental): Bowen's Technique The session lasted for 20 minutes, 3 sessions/week 6th week
  Interventions: Other: Bowen's Technique
- Conventional Physical Therapy (Active Comparator): Conventional Physical Therapy with myofascial release The session lasted for 20 minutes, 3 sessions/week 6th week
  Interventions: Other: Convention Physical Therapy

INTERVENTIONS:
Other: Bowen's Technique — The thumb of the therapist was placed on the top of the targeted muscle (upper trapezius, levator scapulae, tight pectoralis and sternocleidomastoid, longissimus capitis, splenius capitis cervical multifidus). The skin was carried away gently from the spine without disturbing the muscle. The thumb was then hooked into the lateral aspect of the muscle to form a pressure on the muscle. Then the thumb was flattened in the medial direction, when this happened the muscle would plop or 15 respond in some way. Heating pad + TENS will be given The session lasted for 20 minutes 3sessions/week for 6th week
  Arms: Bowen's Technique
Other: Convention Physical Therapy — Myofascial Release + Active Range of Motion Deep transverse friction was given for 10 minutes followed by myofascial stretching of muscle for 3 times, each holding for 90 seconds. Then myofascial release was given using ulnar border of both palms of the therapist.
  Active range of motion exercises will be given 10 reps with 5 seconds hold. Heating pad + Transcutaneous Electrical Nerve Stimulator (TENS) will be given The session lasted for 20 minutes 3sessions/week for 6th week
  Arms: Conventional Physical Therapy

SUMMARY:
No previous randomized control trial has investigated the effectiveness of Bowen's technique on health status in dentists suffering from postural neck Neck pain. Moreover, there is limited evidence and low agreement regarding the effect of Bowen's therapy on Neck pain. Thus, this study aims to answer the question: bowmen's technique is effective for improving Neck pain dentists' function by reducing pain, and disability, and improving posture, and health status, without need for ergonomic alternation?"

DETAILED DESCRIPTION:
Bowen technique may be used for relaxation of tightening muscles in poor posture. The findings suggest that Bowen Therapy has inconsistent immediate effects on postural control and pain threshold in healthy subjects. Further studies are needed using symptomatic participants. No previous randomized control trial, to our knowledge, has investigated the effectiveness of Bowen's technique on health status in dentists suffering from postural neck pain. Moreover, there is limited evidence and low agreement regarding the effect of Bowen's therapy on neck pain. Thus, this study aims to answer the question: Bowen's technique is effective for improving neck pain dentists' function by reducing pain, and disability, and improving posture, and health status, without need for ergonomic alternation?"

ELIGIBILITY:
Inclusion Criteria:

* Both male and females
* Age between 25-50 years. ( House officers and Assistant professor)
* Working hours >5 hours.
* History of cervical pain >2 months.
* Year of practice =<1 year
* Treated more than 5 patient a day

Exclusion Criteria:

* Cervical fracture
* Cervical radiculopathy
* Any surgery to neck and shoulder
* Rheumatoid arthritis
* Sever pain according to Numeric pain rating scale (NPRS)
* Long term anticoagulant or corticosteroid therapy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Modified Goniometer | 6th week
  Modified goniometer can be used to measure craniovertebral angle which is helpful to assess the level of postural disability like forward head posture. It provides an estimation of head on neck angle and position of upper cervical spine.
Numerical Rating Scale | 6th week
  In a Numerical Rating Scale (NRS), patients circle the number between 0 and 10, 0 and 20 or 0 and 100 according to their pain intensity. It is numeric version of visual analog scale.
Neck Disability Index | 6th week
  This is a standard instrument for measuring disability due to neck pain and it's a self-reported questionnaire. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score.

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (4):
- Pakistan (4):
  - Bakhtawar Amin Physiotherapy and Rehabilitation Center, Multan Khurd, Punjab Province
  - Ibn e Sina hospital, Multan Khurd, Punjab Province
  - Nishtar Medical Hospital, Multan Khurd, Punjab Province
  - Salma Medical Center, Multan Khurd, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalal P, Kage V. Comparison Of Ischaemic Compression, Myofascial Release And BowenS Technique In Non Specific Neck Pain-A Randomized Clinical Trial. Indian Journal of Applied Research. 2020;10(1).
- [Background] Nitsure P, Kothari N. THE EFFECTIVENESS OF BOWEN TECHNIQUE AS AN ADJUNCT TO CONVENTIONAL PHYSIOTHERAPY ON PAIN AND FUNCTIONAL OUTCOMES IN SUBJECT WITH ACUTE TRAPEZITIS-A PILOT STUDY. Romanian Journal of Physical Therapy/Revista Romana de Kinetoterapie. 2015;21(36).
- [Background] Al Wazzan KA, Almas K, Al Shethri SE, Al-Qahtani MQ. Back & neck problems among dentists and dental auxiliaries. J Contemp Dent Pract. 2001 Aug 15;2(3):17-30. PMID 12167924
- [Background] Gupta BD, Aggarwal S, Gupta B, Gupta M, Gupta N. Effect of Deep Cervical Flexor Training vs. Conventional Isometric Training on Forward Head Posture, Pain, Neck Disability Index In Dentists Suffering from Chronic Neck Pain. J Clin Diagn Res. 2013 Oct;7(10):2261-4. doi: 10.7860/JCDR/2013/6072.3487. Epub 2013 Oct 5. PMID 24298492
- [Background] Abiodun-Solanke IM, Agbaje JO, Ajayi DM, Arotiba JT. Prevalence of neck and back pain among dentists and dental auxiliaries in South-western Nigeria. Afr J Med Med Sci. 2010 Jun;39(2):137-42. PMID 21117410
- [Background] Letafatkar A, Rabiei P, Alamooti G, Bertozzi L, Farivar N, Afshari M. Effect of therapeutic exercise routine on pain, disability, posture, and health status in dentists with chronic neck pain: a randomized controlled trial. Int Arch Occup Environ Health. 2020 Apr;93(3):281-290. doi: 10.1007/s00420-019-01480-x. Epub 2019 Oct 25. PMID 31654125
- [Background] Pargali N, Jowkar N. Prevalence of musculoskeletal pain among dentists in Shiraz, Southern Iran. Int J Occup Environ Med. 2010 Apr;1(2):69-74. PMID 23022788